CLINICAL TRIAL: NCT04824625
Title: Observational Study of the Incidence of Infection Reported by SARS CoV-2 in Attendees of a Commercial Music Concert at the Palau Sant Jordi (Barcelona)
Brief Title: Incidence of Infection Reported by COVID-19 in Attendees of a Commercial Music Concert
Status: Completed | Type: Observational
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Festivals per la Cultura Segura AIE (Unknown)
Responsible Party: Sponsor
Other Study IDs: StJordi-CoV
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Covid-19 (SARS-CoV-2)
Keywords: SARS-CoV-2; COVID-19; Coronavirus; Superspreading event; Concert
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
From the beginning of the pandemic caused by SARS-CoV-2, most events with massive participants have been canceled due to being considered high-risk events for the SARS-CoV-2 transmission. It has been detected that asymptomatic people infected by SARS-CoV-2, are playing an important role in the contagious in these kinds of events. The economic losses arising from the closure of these activities, mainly those related to culture and musical performances are around 2.5 billion euros a Catalonia, and a considerable loss of jobs in this sector.

Developing strategies of cribrate of infected people by SARS-CoV-2 asymptomatic or not diagnosticated and with a potential transmission of the virus is the key to perform cultural, sport, etc. massive events with all the security. The objective is to exclude infected people with a a high potential of transmission.

It is needed to use versatile tests for this objective, so the test must have a high sensibility to detect infected people, the test has to be easy to manipulate without requiring a high technology of the laboratory hospitals, neither prolongated to obtain a result and that has a low cost. The rapid SARS-CoV-2 antigen screening tests are best suited for this purpose.

On 27th March, a musical concert will be performed at Palau St Jordi (Barcelona) with 5000 attendees and with all the SARS-COV-2 safety measures by the "Secretary General of Health of the Generalitat de Catalunya" a (mandatory wearing a mask during the event, restricted outdoor areas of bar and smoking enhanced ventilation of the whole indoor area and avoiding queues.). This study wants to assess the incidence of SARS-CoV-2 infection reported to the health system among the attendees of this commercial concert during the 14 days following the event, also it will be evaluated the clinical evolution of the possible infections during the concert.

DETAILED DESCRIPTION:
From the beginning of the pandemic caused by SARS-CoV-2, most events with massive participants have been canceled due to being considered high-risk events for the SARS-CoV-2 transmission. It has been detected that asymptomatic people infected by SARS-CoV-2, are playing an important role in the contagious in these kinds of events. The economic losses arising from the closure of these activities, mainly those related to culture and musical performances are around 2.5 billion euros a Catalonia, and a considerable loss of jobs in this sector.

Developing strategies of cribrate of infected people by SARS-CoV-2 asymptomatic or not diagnosticated and with a potential transmission of the virus is the key to perform cultural, sport, etc. massive events with all the security. The objective is to exclude infected people with a a high potential of transmission.

It is needed to use versatile tests for this objective, so the test must have a high sensibility to detect infected people, the test has to be easy to manipulate without requiring a high technology of the laboratory hospitals, neither prolongated to obtain a result and that has a low cost. The rapid SARS-CoV-2 antigen screening tests are best suited for this purpose. These tests have shown a sensitivity close to 99% to detect infectious people who have a high viral load of SARS-CoV-2. No viral isolation has been demonstrated in any culture of samples of patients infected with SARS-CoV-2 with a Ct threshold (cycle threshold) in the test RT-PCR greater than 30, which is considered to delimit the transmitting potential of the infected

On 27th March, a musical concert will be performed at Palau St Jordi (Barcelona) with 5000 attendees and with all the SARS-COV-2 safety measures by the Secretaria General de Salut de la Generalitat de Catalunya (mandatory wearing a mask during the event, restricted outdoor areas of bar and smoking enhanced ventilation of the whole indoor area and avoiding queues.). This study wants to assess the incidence of SARS-CoV-2 infection reported to the health system among the attendees of this commercial concert during the 14 days following the event, also it will be evaluated the clinical evolution of the possible infections during the concert.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years and under 65) attending the commercial music event scheduled at the Palau Sant Jordi
* Sign informed consent, including an authorization for the collection of data from the electronic health system of the Catalan System of Health on the notification of COVID-19 infection during the 14 days following the event or authorization to be contacted by telephone by the medical team, if necessary, for complete information on SARS-CoV-2 infection.

Exclusion Criteria:

* Minors (<18 years)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the commercial concert attendees, that are major of age (>18 years old) and who have signed the informed consent to access their Medical records 14 days after the commercial concert.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2021-03-27 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Incidence rate of people with SARS-CoV-2 | From day 1 to day 14 after the event
  Incidence rate of assistants with reported SARS-COV-2 14 dys after the event
Incidence rate of consultations in primary care centers | From day 1 to day 14 after the event
  Incidence rate of consultations in primary care centers about symptoms compatible with COVID-19 during the 14 days after the event

SECONDARY OUTCOMES:
Incidence rate of Hospital emergencies | From day 1 to day 14 after the event
  Incidence rate of hospital emergencies about symptoms compatible with COVID-19 during the 14 days after the event
Incidence rate of hospital admissions | From day 1 to day 14 after the event
  Incidence rate of hospital admissions about symptoms compatible with COVID-19 during the 14 days after the event
Incidence rate of Intensive care units admissions | From day 1 to day 14 after the event
  Incidence rate of intensive care units in the concert participants with COVID-19 during the 14 days after the event
Incidence rate of mortality | From day 1 to day 14 after the event
  Incidence rate of COVID-19 mortality in the concert participants during the 14 days after the event

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain